CLINICAL TRIAL: NCT02609555
Title: Trans-anal Endoscopic Microsurgery (TEM) Assisted Perineal Rectopexy With Postanal Repair and Anal Cerclage In Treatment of Rectal Prolapse (Novel Technique)
Brief Title: TEM Assisted Perineal Rectopexy in Treatment of Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MansouraU26
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Rectal Prolapse
Keywords: TEM; Rectopexy; rectal prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TEM perineal Rectopexy (Experimental): TEM perineal rectopexy: triple repair technique , Perineal rectopexy with a polyprolene mesh assisted by TEM technique, postanal repair to close the postanak space then finally anal cerclage to hold the rectum in place for one month.
  Interventions: Procedure: TEM perineal rectopexy

INTERVENTIONS:
Procedure: TEM perineal rectopexy — perineal rectopexy using polyprolene mesh assisted by TEM technique and special proctoscope postanal repair in two layers to narrow the postanal space anal cerclage with absorbable sutures

SUMMARY:
Curvilinear incision in the postanal space, through the intersphincteric plane, insertion of Proctoscope of TEM technique and dissection till sacral promontory, insertion of mesh between the rectum and sacrum, post anal repair then anal cerclage width absorbable suture.

DETAILED DESCRIPTION:
Perineal Rectopexy is performed by an incision in the intersphincteric space followed by dissection till the sacral promontory then Proctoscope is inserted to complete the dissection .Mesh is inserted and fixed to the sacrum with laparoscopic tacker ( or can be left unfixed) then postanal repair is conducted in two layers ( levatorplasty then sphincteroplasty) and finally Ana cerclage is done with polyglactin 0 sutures

ELIGIBILITY:
Inclusion Criteria:

* patients with complete or partial rectal prolapse

Exclusion Criteria:

* patients unfit for surgery
* patients with previous surgery for rectal prolapse
* patients with associated anorectal pathology (e.g fistula )
* patients with constipation as a predominant symptom.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of prolapse | 12 months
  Number of patients presenting with recurrent rectal prolapse within 12 months after surgery

SECONDARY OUTCOMES:
Improvement of continence state | 12 months
  Amount of increase in continence score after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt